CLINICAL TRIAL: NCT02124642
Title: Folic Acid Supplementation in Pregnant Women: Dose Response
Acronym: FAPREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: University of Florida (Other); Emory University (Other); Cornell University (Other)
Responsible Party: Principal Investigator, Lynn B. Bailey, PhD, Department Head and Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: FASUPPPREG-2014
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy
Keywords: Folate requirements; Pregnancy; Folic acid; DNA methylation; Folate biomarkers
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folic acid, 400 mcg/day (Active Comparator): A daily 400 microgram (mcg) dose of folic acid will be taken orally, along with the recommended intake for pregnancy of other vitamins, minerals and docosahexaenoic acid (DHA), beginning at enrollment until delivery. The 400 mcg dose approximates the current Recommended Dietary Allowance (RDA) for pregnant women of 600 mcg Dietary Folate Equivalents (400 mcg folic acid ≈ 600 mcg DFEs; conversion factor based on higher bioavailability of folic acid is: 1 mcg folic acid = 1.7 mcg DFE).
  Interventions: Dietary Supplement: Folic acid, 400 mcg/day
- Folic acid, 800 mcg/day (Experimental): A daily 800 microgram (mcg) dose of folic acid will be taken orally, along with the recommended intake for pregnancy of other vitamins, minerals and docosahexaenoic acid (DHA), beginning at enrollment until delivery. The 800 microgram dose, which is considerably higher than the current RDA, represents an amount commonly found in over-the-counter prenatal vitamin formulations.
  Interventions: Dietary Supplement: Folic acid 800 mcg/day

INTERVENTIONS:
Dietary Supplement: Folic acid, 400 mcg/day — The supplement regime for this arm will consist of (1) a women's multivitamin/ multimineral (MVM) supplement containing 400 mcg folic acid, (2) a capsule containing 200 mg DHA and (3) a capsule formulated to contain 10 mg iron (which represents the difference in the amount of iron in the women's MVM formulation and that in prenatal MVM supplements).
  Arms: Folic acid, 400 mcg/day
Dietary Supplement: Folic acid 800 mcg/day — The supplement regime for this arm will consist of (1) a women's multivitamin/ multimineral (MVM) supplement containing 400 mcg folic acid, (2) a capsule containing 200 mg DHA and (3) a capsule formulated to contain 10 mg iron (which represents the difference in the amount of iron in the women's MVM formulation and that in prenatal MVM supplements) and 400 mcg folic acid.
  Arms: Folic acid, 800 mcg/day

SUMMARY:
The proposed study is a double-blind randomized controlled trial in healthy pregnant women (BMI 18.5 - 29.9 kg/m2, age 18 - 40 yr) receiving prenatal care at Athens Regional Midwifery clinic (ARMC).

The primary goal of the proposed study is to determine relative changes in blood folate and DNA methylation levels in response to 2 different supplemental doses of folic acid one of which will provide the Institute of Medicine's recommended folate intake for pregnant women and the second will provide a higher dose as routinely taken by pregnant women in over-the-counter prenatal supplements.

The specific aims of the study are:

1. to compare maternal serum and red blood cell (RBC) folate levels and % change in women taking either 400 or 800 mcg/day of supplemental folic acid from the first prenatal visit (< 10 weeks) through delivery;
2. to compare the infant's cord blood folate levels in response to different maternal folic acid intakes (400 mcg/d vs 800 mcg/d);
3. to determine relative differences in the levels of oxidized folic acid in maternal and infant blood in response to 400 or 800 mcg/d folic acid dose, and
4. to determine genome wide and gene specific DNA methylation response in pregnant women receiving prenatal supplements containing either 400 or 800 mcg folic acid per day

DETAILED DESCRIPTION:
The study will be conducted in healthy women with a BMI within the ranges of 18.5 - 35.0 kg/m2. There will be two treatment groups: (1) one group taking 400 mcg per day of folic acid as part of a prenatal supplement, beginning at study enrollment (< 10 weeks gestational age) and (2) a second group taking 800 mcg per day of folic acid as part of the prenatal supplement. Both groups will be provided identical composition of prenatal supplements other than folic acid content. Repeated measures of outcome variables will be determined in blood samples collected at various times during pregnancy and at delivery. Due to the role of prenatal supplementation in helping maintain optimal nutrition status throughout pregnancy, there will be no placebo control.

Women will be recruited through the Athens Regional Medical Center Midwifery Practice and all blood draws associated with this study will be conducted during scheduled prenatal visits. The research protocol is consistent with the standard of care provided by the clinic and will not affect the prenatal services provided to the research participants. Following consent at the first prenatal visit, participants will be randomly assigned to receive prenatal supplements containing either 400 or 800 mcg of folic acid (all other ingredients at unmodified concentrations). The 400 mcg dose approximates the current Recommended Dietary Allowance (RDA) for pregnant women of 600 mcg Dietary Folate Equivalents (400 mcg folic acid ≈ 600 mcg DFEs; conversion factor based on higher bioavailability of folic acid is: 1 mcg folic acid = 1.7 mcg DFE). The higher dose of 800 mcg folic acid represents an amount commonly found in over-the-counter prenatal supplements. Women will be asked to take the supplements daily throughout the duration of gestation and to follow their standard prenatal diet, with the exception of avoiding highly fortified (> 100% RDA) ready-to-eat cereals and fortified energy/snack bars and drinks, due to their high folic acid content.

At the first visit, the participants will be instructed in the use of a dietary recall data collection sheet (food diary) which they will be asked to complete during specific time points during the study. Each set of dietary recalls will include information for three 24-hr periods on non-consecutive days including one weekend day. Dietary recall information will be obtained at approximately weeks 16 and 32 of gestation. This will permit assessment of typical dietary intake of total calories and specific nutrients, including folate.

Blood samples will be collected, in the non-fasting state, at the first, 28 week and 36 week prenatal visits and from the mother and cord blood at delivery for determination of primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women with singleton pregnancy
* < 10 weeks gestation at enrollment
* body mass index 18.5 - 35.0 kg/m2
* willingness to comply with study protocol ( i.e. take assigned daily prenatal vitamin; complete diet recall and study questionnaire)
* not consuming super-fortified ready-to-eat cereal products (with > 100% RDA for folate per serving)

Exclusion Criteria:

* BMI < 18.5 or > 35.0 kg/m2
* use of prescription drugs
* anemia
* chronic disease (diabetes, hypertension, epilepsy, cancer, kidney disease, cardiovascular disease)
* acute illness (e.g. pneumonia, urinary tract infection, mononucleosis)
* use of antibiotics in past 2 weeks
* follows vegan dietary regime
* current smoker
* typical alcohol consumption of 2 or more drinks per day
* having undergone in vitro fertilization treatment
* carrying more than one fetus
* pregnancy-associated complications (i.e gestational diabetes, pre-eclampsia)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum folate | Baseline (Initial Prenatal Visit), 28 and 36 weeks gestation, delivery
  Change in serum folate concentrations in response to supplementation during pregnancy with one of two levels of folic acid will be determined by microbiological assay using Lactobacillus rhamnosus. Cord blood serum folate at delivery will also be determined by the microbiological assay. Differences in serum folate response to the two levels of folic acid supplementation will be compared.
Red blood cell (RBC) folate | Baseline (Initial Prenatal Visit), 28 and 36 weeks gestation, delivery
  Change in red blood cell (RBC) folate concentrations in response to supplementation during pregnancy with one of two levels of folic acid will be determined by microbiological assay using Lactobacillus rhamnosus. Cord blood RBC folate at delivery will also be determined by the microbiological assay. Differences in RBC folate response to the two levels of folic acid supplementation will be compared.
Serum folic acid | Baseline (Initial Prenatal Visit), 28 and 36 weeks gestation, delivery
  Change in serum folic acid concentrations in response to supplementation during pregnancy with one of two levels of folic acid will be determined by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Cord blood serum folic acid at delivery will also be determined by LC-MS/MS. Differences in serum folic acid in response to the two levels of folic acid supplementation will be compared.
Gene-specific DNA methylation | Baseline (Initial Prenatal Visit), 28 and 36 weeks gestation, delivery
  Change in DNA methylation in response to folic acid supplementation during pregnancy will be determined in DNA isolated from whole blood. Illumina Infinium HumanMethylatio450 bead chip microarrays will be used to assess changes in multiple methylation sites of specific genes within regulatory pathways for folate metabolism and/or development. Differences in DNA methylation in response to the two levels of folic acid supplementation will be compared.
  We anticipate analyzing DNA methylation response at multiple time points and in all participants. Due to the expense associated with the analysis, however, we may be able to perform the analysis only at baseline and delivery and in only a subset of the participants if we are unable to secure additional funding.

SECONDARY OUTCOMES:
Cell-type-specific DNA methylation | Baseline (Initial Prenatal Visit), 28 and 36 weeks gestation, delivery
  Change in DNA methylation in response to folic acid supplementation during pregnancy will be determined in DNA isolated from specific white blood cell types obtained by antibody/magnetic technology. Illumina Infinium HumanMethylatio450 bead chip microarrays will be used to assess changes in multiple methylation sites of specific genes within regulatory pathways for folate metabolism and/or development. Differences in DNA methylation in response to the two levels of folic acid supplementation will be compared.
Infant birth weight | Delivery
  Birth weight information will be obtained from medical records
Infant length | Delivery
  Length at birth will be obtained from medical records
Infant head circumference | Delivery
  Infant head circumference will be obtained from medical records.
Apgar score | Delivery
  Apgar score of the infant will be obtained from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn B Bailey, PhD, Principal Investigator — University of Georgia; Dorothy B Hausman, PhD, Study Director — University of Georgia; Hea Jin Park, PhD, Study Director — University of Georgia; Gail P A Kauwell, PhD, RDN, Study Director — University of Florida; Marie A Caudill, PhD, RD, Study Director — Cornell University; Alicia K Smith, PhD, Study Director — Emory Univeristy
Locations (1):
- Athens Regional Medical Center Midwifery Practice, Athens, Georgia, United States